CLINICAL TRIAL: NCT00088777
Title: Behavioral Preparation for Treating Fibromyalgia
Brief Title: Nondrug Treatment Programs for Adults With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Akiko Okifuji, University of utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9345; 5R01AR048888-06 (NIH); R01AR048888-01A2 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- MET (Experimental)
  Interventions: Behavioral: Behavioral coping skills training plus physical therapy
- CSE (Experimental)
  Interventions: Behavioral: Stress management education plus physical therapy

INTERVENTIONS:
Behavioral: Behavioral coping skills training plus physical therapy — 10 hours coping sessions, 6 hours activating physical therapy, 4 hours physical therapy education
  Arms: MET
Behavioral: Stress management education plus physical therapy — 10 hours stress management education, 6 hours activating physical therapy, 4 hours physical therapy education
  Arms: CSE

SUMMARY:
Fibromyalgia (FM) syndrome is a common chronic pain disorder that may benefit from nondrug treatment. This study will compare the effectiveness of behavioral preparation, stress management education, and fibromyalgia and coping education in relieving the symptoms of FM. Each of these nondrug treatments will be combined with physical therapy and physical education.

Specific aims: 1) Evaluate the efficacy of behavioral preparation programs on attrition, compliance, and treatment outcomes of self-management rehabilitation for FM syndrome. 2) Determine factors that mediate clinical efficacy. 3) Evaluate individual differences in treatment responses to delineate who will benefit most from each type of the behavioral preparation programs.

DETAILED DESCRIPTION:
FM is a chronic pain condition causing discomfort and disability; there is no known cure. Research suggests that combination treatment of physical therapy, fibromyalgia education, and stress management education is helpful for many patients with this condition. However, how much benefit patients get from such therapies varies greatly. This study will evaluate the effectiveness of behavioral preparation, stress management education, and fibromyalgia and coping education each in combination with physical therapy and physical education, in relieving the symptoms of FM.

The study will last approximately 15 months. Participants will undergo a comprehensive assessment including medical, physical, and psychological evaluations. Blood will be collected to measure participants' serotonin levels; participants will also be asked to complete several questionnaires to assess their FM symptoms and joint function. For a 7-day period prior to starting behavioral interventions, participants will be asked to carry a personal-size digit assistant (PDA) that will ask them questions about their quality of life three times a day . During this time, they will also continuously wear a wristwatch-like device to measure functional movement and quality of sleep.

For 10 weeks, participants will undergo therapy sessions of one of the behavioral interventions (behavioral preparation, stress management education, or fibromyalgia and coping education) along with physical therapy and physical education. During Weeks 1 through 4, participants will receive 2 hours of their assigned intervention. During Weeks 5 and 6, they will receive 1 hour of their assigned intervention and 1 hour of physical therapy. During Weeks 7 through 9, they will receive 1 hour of physical therapy and 1 hour of physical education. During Week 10, they will receive 1 hour of their assigned intervention and 1 hour of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* Have not been actively exercising (e.g., aerobic activity such as cycling, jogging, climbing, rowing, and muscle strengthening activity) for more than 30 minutes per week

Exclusion Criteria:

* Other progressive disease
* Plan to have surgery during the next year
* Pregnancy or planning to become pregnant during the next year
* Resting diastolic blood pressure greater than 115 mm Hg or resting systolic blood pressure greater than 200 mg Hg
* Cardiovascular diseases
* Serious psychopathology (e.g., diagnoses of psychosis, organic mental disorder, or dissociative disorder; active suicidal intent; inpatient admission to psychiatric ward or incidence of self-injurious behaviors in the past year)
* Non-IV substance abuse within the last 2 years, or history of recreational IV drug use
* Other rheumatologic disorder (e.g., rheumatoid arthritis)
* Neuropathic pain
* Pain associated with terminal illness, acute pain, or pain associated with specific organ damage (e.g., stomach ulcer)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Major FM syndrome symptoms immediately following treatment and at 6- and 12-month follow-up evaluations | post-treatment, 6 month and 12 month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Okifuji, PhD, Principal Investigator — University of Utah, Pain Research and Management Center
Locations (1):
- University of Utah, Pain Research and Management Center, Salt Lake City, Utah, United States